CLINICAL TRIAL: NCT00756314
Title: Effectiveness of Contraceptive Counseling of Women Following an Abortion in Recife, Brasil: a Randomized Controlled Intervention Study.
Brief Title: Contraceptive Counseling Following an Abortion
Acronym: APA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Materno Infantil Prof. Fernando Figueira (Other)
Responsible Party: Ana Laura Carneiro Gomes Ferreira, IMIP
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: APA-1
Record Dates: First submitted 2008-09-19; First posted 2008-09-22 (Estimated); Results first posted 2010-09-30 (Estimated); Last update posted 2010-10-13 (Estimated); Status verified 2010-03

CONDITIONS: Post Abortion Care
Keywords: Ambulatory Care Facilities; abortion care; contraception; counseling; outpatient clinic
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Personalized contraceptive counseling (Experimental): All 123 allocated women for the intervention group received personalized counseling (face-to-face) and the contraceptive method chosen for free by a specialized trained doctor in family planning.
  Interventions: Behavioral: Personalized contraceptive counseling
- Control (No Intervention): All 123 women allocated to control group received a standard care available at IMIP.Standard care is comprised of educational group counseling by specialized nursing staff in family planning discussing about contraceptive methods and side effects
  Interventions: Behavioral: Personalized contraceptive counseling

INTERVENTIONS:
Behavioral: Personalized contraceptive counseling — The intervention comprised a personalized and comprehensive (face-to-face) contraceptive counseling regarding to individual contraceptive history and needs. The counseling intervention was conducted by three trained gynecologists according to standard one day training.
  Other Names: Intervention group; Control group

SUMMARY:
The purpose of this study is to determine whether contraceptive counseling is effective on acceptance and use of methods in women following an abortion.

DETAILED DESCRIPTION:
Contraceptive counseling is considered an essential component of post abortion care (PAC) programmes and it is recommended to prevent unintended pregnancies and unsafe, repeated abortions. Indeed, most maternal deaths related to unsafe abortions could be prevented by expanding and improving family planning provision.

ELIGIBILITY:
Inclusion Criteria:

* Within the first 10 days (plus or minus 5 days) after an abortion
* Live in Recife or whereabouts in Recife(Brazil)

Exclusion Criteria:

* Clinical diagnosis of Gestational Trophoblastic Disease
* Women HIV positive
* Psychiatric pathology

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 246 (Actual)
Dates: Start 2008-07; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ariani I Souza, PhD, Study Director — IMIP
Locations (1):
- IMIP - Instituto Materno Infantil Prof Fernando Figueira, Recife, Pernambuco, Brazil

REFERENCES:
- See also: Click here for more information about the study location (sponsor) — http://www.imip.org.br

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period was between July 2008 and September 2009. All women who had an abortion in any of the five public maternities in Recife were invited to participate.
Pre-assignment Details: Of the 403 women invited, 310 attended the service. However 39 women were excluded because they did not agree to participate and 25 women did not fill the inclusion criteria, as for gestational trophoblastic disease, benign and malignant tumors of the uterus and uterine malformation.
Groups:
- Personalized Contraceptive Counseling: All allocated women for the intervention group received personalized counseling (face-to-face) and the contraceptive method chosen for free by a specialized trained doctor in family planning.
- Control: All women allocated to control group received a standard care available at IMIP.Standard care is comprised of educational group counseling by specialized nursing staff in family planning discussing about contraceptive methods and side effects
Period: Overall Study
Arm/Group | Personalized Contraceptive Counseling | Control
Started | 123 | 123
Completed | 121 (2 participants discontinued the intervention and were analyzed by "intention to treat" analysis.) | 64 (4 participants did not do the follow up, 55 discontinued and were analyzed by "intention to treat")
Not Completed | 2 | 59
Not completed — Lost to Follow-up | 2 | 59

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Personalized Contraceptive Counseling | Control | Total
Number analyzed (Participants) | 123 | 123 | 246
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11 | 8 | 19
  Between 18 and 65 years | 112 | 115 | 227
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 26.2 (6.8) | 27.6 (6.8) | 26.6 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 123 | 123 | 246
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Brazil | 123 | 123 | 246

OUTCOME MEASURES:

1. Primary Outcome: Contraceptive Acceptability and Use of Contraceptives During the 6-month Follow-up
Description: The acceptability and the use of contraceptives during the follow-up period was defined as just "yes" or "no"
Time Frame: after the contraceptive counseling and during the 6-month follow
Population: The analysis was by "intention to treat" in both groups. All the women were retained in their original assigned group.
Measure: Number; unit: participants
Units Other Than Participants: participants
Arm/Group | Personalized Contraceptive Counseling | Control
Number analyzed (Participants) | 123 | 123
participants | 121 | 86

2. Primary Outcome: Correct Use of the Method
Description: the correct use was considerer by each methods according the prescription.
Time Frame: within the first 6 months after intervention
Measure: Number; unit: participants
Arm/Group | Personalized Contraceptive Counseling | Control
Number analyzed (Participants) | 123 | 123
participants | 121 | 68

3. Secondary Outcome: Pregnancies Among All Women
Time Frame: within the first six months after intervention
Measure: Number; unit: participants
Arm/Group | Personalized Contraceptive Counseling | Control
Number analyzed (Participants) | 123 | 123
participants | 2 | 12

4. Primary Outcome: Chosen Contraceptive Method After Counseling
Description: the type of contraceptive methods chosen by women following after counseling
Time Frame: after the contraceptive counseling
Measure: Number; unit: participants
Arm/Group | Personalized Contraceptive Counseling | Control
Number analyzed (Participants) | 123 | 123
participants | 123 | 117

5. Secondary Outcome: Satisfaction With the Used Contraceptive Method
Description: the satisfaction was measured according a scale ranging in 3 levels: very satisfied, somewhat satisfied and dissastisfied.
Time Frame: During the 6-month Follow-up
Measure: Number; unit: participants
Arm/Group | Personalized Contraceptive Counseling | Control
Number analyzed (Participants) | 123 | 123
participants | 99 | 41

ADVERSE EVENTS:
Time Frame: nausea and vomiting with use of the pill, one of the methods prescribed
Arm/Group | Personalized Contraceptive Counseling | Control
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/48
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The time of the follow up of six months after the abortion, not having the possibility to evaluate the effectiveness of the measurement in longer term.

However, this decision may have contributed to overestimate the intervention effect.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes